CLINICAL TRIAL: NCT05066074
Title: Comparison of the Safety and Efficacy Between the Distal and Proximal Radial Vascular Access Technique in Coronary Diagnostic and Therapeutic Procedures
Brief Title: Safety and Efficacy Between the Distal and Proximal Radial Vascular Access Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Manuel Alonso Abril Lee, Interventional Cardiology Consultant, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17 C102 004 049
Record Dates: First submitted 2021-09-14; First posted 2021-10-04 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Coronary Artery Disease
Keywords: radial artery; distal radial artery; vascular access; radial artery occlusion
MeSH Terms: conditions — Coronary Artery Disease; Arterial Occlusive Diseases

STUDY DESIGN:
Intervention Model Description: Randomised Clinical Trial - Equivalence model (Two tailed) Based on a previous pilot study: SD 97 sec Allowable Diff: 90 sec, Patient loss 15%, Type I error 2.5%, Type II error 90% Mean Differences: 0
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Distal Radial Access (Experimental): Distal Radial (Anatomical Snuffbox) Vascular Access prior to catheterization
  Interventions: Procedure: Distal Radial Vascular Access
- Proximal Radial Access (Active Comparator): Proximal Radial Vascular Access prior to catheterization
  Interventions: Procedure: Distal Radial Vascular Access

INTERVENTIONS:
Procedure: Distal Radial Vascular Access — Distal Radial Vascular Access
  Other Names: dTRA

SUMMARY:
The investigators are conducting a randomized clinical trial, having as a primary objective, to compare vascular access time between distal and proximal radial approach. Secondary objectives include comparing incidence of distal and proximal radial artery occlusion, at 24 hrs and 30 days. As a tertiary objective investigators will compare the preference of the patients for each access in subsecuent interventional procedures.

DETAILED DESCRIPTION:
Randomised Clinical Trial / Equivalence Model Permutted block asignation 1:1 Statistical Power 90% and Significance 2.5%. Sample Loss estimation - 15% Chi-square to categorical and T Student to numerical variables. Logistic regression binomial for adverse outcomes. If needed, an intention to treat analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Clinical indication for coronary angiography / angioplasty
* Palpable radial and distal radial pulse
* Previous clinical Barbeau test
* Radial and distal radial patency via vascular ultrasound
* 24-hour and 30-day follow-up feasibility

Exclusion Criteria:

* Previous vascular punctions in the studied anatomic site
* Artery introductor relationship
* Arteriovenous fistula
* Current treatment with oral anticoagulants
* Contraindication for Heparin
* Incomplete medical records
* Vascular access sheath - radial artery mismatch
* Distal radial or ulnar fracture history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-08-16 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Vascular Access Time | Seconds during the procedure
  Starts when the anesthesia needle contacts the skin and stops when the introducer sheath has been properly placed and flushed.

SECONDARY OUTCOMES:
"Conventional" Radial Artery Occlusion | In the first 24 hours, and follow up to 30 days
  Radial Artery Occlusion using vascular ultrasound
Distal Radial Artery Occlusion | In the first 24 hours, and follow up to 30 days
  Distal Radial Artery Occlusion using vascular ultrasound

OTHER OUTCOMES:
Quality of life outcome | 30-day survey
  Patient preference for the same access in case a second procedure is needed

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Mexicano del Seguro Social, Tijuana, Estado de Baja California, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: (planned) March 2022